CLINICAL TRIAL: NCT01653639
Title: Single Dose, Open-label, Randomized, Crossover Study in Subjects With Severe Hemophilia A to Compare the Bioavailability of 2 Different Strengths of Kogenate FS (BAY14-2222)
Brief Title: Comparative Pharmacokinetic Study of Two Different Strengths of BAY14-2222
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15495; 2012-001045-40 (EudraCT Number)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Hemophilia A
Keywords: BAY14-2222; Pharmacokinetics
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)
- Arm 2 (Experimental)
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — 50 IU/kg single dose using the 3000 IU vial size (600 IU/ml)
  Arms: Arm 1
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — 50 IU/kg single dose using the 2000 IU vial size (400 IU/ml)
  Arms: Arm 2

SUMMARY:
This is a single dose, open-label, randomized, crossover study in subjects with severe Hemophilia A to compare the bioavailability of 2 different strengths of Kogenate FS (BAY 14-2222).

ELIGIBILITY:
Inclusion Criteria:

* Males, age 18 to 65 years
* Subjects with Severe hemophilia A with a documented plasma FVIII level of <1%
* >/= 150 ED (exposure days) with FVIII concentrates(s) as supported by medical records

Exclusion Criteria:

* Evidence of current or past inhibitor antibody
* History of any congenital or acquired coagulation disorders other than hemophilia A
* Platelet count <75,000/mm3
* Abnormal renal function (serum creatinine >2 times the upper limit of the normal range)
* Active liver disease verified by medical history or persistently elevated alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5x the upper limit of normal or severe liver disease as evidenced by, but not limited to any of the following: International Normalized Ratio (INR) >1.4, hypoalbuminemia, portal vein hypertension including presence of otherwise unexplained splenomegaly and history of esophageal varices

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of BAY14-2222 | Up to 48 hours
Area under the plasma concentration vs time curve from time 0 to time of last measurable concentration AUC(0-tlast) of BAY14-2222 | Up to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Sofia, Bulgaria